CLINICAL TRIAL: NCT05940792
Title: Immediate Effect of Non-Elastic Taping on Gait Balance in Stroke Patients: Randomized Controlled Trial
Brief Title: Immediate Effect of Non-Elastic Taping on Gait Balance in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Beyzanur Dikmen, Research Assistant, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UskudarU1
Record Dates: First submitted 2023-06-20; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Stroke
Keywords: balance; gait; immediate; stroke; taping
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group received 45 min of conventional physiotherapy after nonelastic taping, which provides eversion support.
  Interventions: Other: Nonelastic taping
- control group (Active Comparator): The control group received 45 min of conventional physiotherapy
  Interventions: Other: Conservative physiotherapy

INTERVENTIONS:
Other: Nonelastic taping — Non-elastic taping was placed on the ankle of the affected side with a plaster band starting from the middle of the sole of the foot and extending from the lateral side of the foot to the level below the knee to provide eversion support.
  Arms: intervention group
Other: Conservative physiotherapy — The conventional physiotherapy programme included range of motion exercises, balance and gait training and neuromuscular electrical stimulation.
  Arms: control group

SUMMARY:
After a stroke, most patients have poor ankle control and difficulty walking. Considering that proper foot placement will provide a more balanced and controlled gait, the aim of this study was to investigate the immediate effect of non-elastic ankle taping providing eversion support on gait balance in stroke patients.

DETAILED DESCRIPTION:
The study included 30 stroke patients. Participants were randomly assigned to two groups: intervention group(n=15) and the control group(n=15). The control group received 45 min of conventional physiotherapy. The intervention group received 45 min of conventional physiotherapy after nonelastic taping, which provides eversion support. The gait balance of both groups was evaluated using the Dynamic Gait Index before and after treatment. . Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* having a stroke diagnosis at least 6 months ago,
* being between the ages of 18 and 75,
* having a spasticity grade of 0, 1, 1+, 2 according to the Modified Ashworth Scale,
* having no cooperation problems and being mobilized without support.

Exclusion Criteria:

* orthopedic problems such as surgical intervention, fracture history, presence of cognitive, visual, or cardiovascular diseases
* skin sensitivity in the foot and ankle that may affect gait.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index (DGI) | 5 months
  The dynamic gait index includes 8 items: walking, walking at different speeds, crossing an obstacle, walking around an obstacle, suddenly turning 180 degrees while walking and stopping, climbing steps, walking by turning the head left and right in the horizontal plane, and walking by turning the head up and down in the vertical plane. The performance of each item was graded with 4 points. The score scale is as follows; 3 independent walking, 2 mild impairment, 1 moderate impairment and 0 severe impairment; the total score that can be obtained varies between 0-24 points. If the total score is between 22and24, it can be said that individuals have safe ambulation, 20-21 points are considered to be a harbinger of fall risk, and scores of 19 or lower have been associated with an increased incidence of falls

CONTACTS AND LOCATIONS:
Overall Officials: Beyzanur Dikmen Hoşbaş, Principal Investigator — Uskudar University; Berna Karamancıoglu, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No